CLINICAL TRIAL: NCT02295852
Title: Effects of Changes in Calcium Dietary Intake on Blood Pressure and Body Weight Control
Brief Title: Increasing Calcium Dietary Intake Helps to Control Blood Presure and Body Weight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Ferrara Liberato Aldo, Associate Professor of Medicine, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2014-11-07; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Hypertension; Body Weight
Keywords: Low-sodium calcium enriched diet; Low-sodium diet; Glucose and lipid metabolims
MeSH Terms: conditions — Hypertension; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: LOW-SODIUM LOW LIPID CALCIUM RICH DIET (Experimental): Experimental Group A: patients will change their diet in a diet similar for total daily calories, sodium and macronutrients but enriched in calcium (1200 mg/daily) and will be followed up to 1 year with an intermediate control after the first 3 months;
  Interventions: Dietary Supplement: LOW-SODIUM LOW LIPID CALCIUM RICH DIET
- Group B: LOW-SODIUM LOW LIPID DIET (Active Comparator): Experimental Group B: patients will continue the low-lipid, low-sodium diet up to 1 year with an intermediate control after the first 3 months.
  Interventions: Dietary Supplement: LOW-SODIUM LOW LIPID DIET

INTERVENTIONS:
Dietary Supplement: LOW-SODIUM LOW LIPID CALCIUM RICH DIET — 1.Composition of the diet: Proteins 17%, Total lipids 28%, Saturated Fatty Acids 7%, Carbohydrates 54%, Fibers 42 g, Sodium 1377 mg, potassium 4067mg, Calcium 1211 mg
  Arms: Group A: LOW-SODIUM LOW LIPID CALCIUM RICH DIET
Dietary Supplement: LOW-SODIUM LOW LIPID DIET — 2. Composition of the diet: Proteins 17%, Total lipids 27%, Saturated Fatty Acids 7%, Carbohydrates 56%, Fibers 39 g, Sodium 1397 mg, potassium 3973 mg, Calcium 650 mg
  Arms: Group B: LOW-SODIUM LOW LIPID DIET

SUMMARY:
Mediterranean diet is relatively poor in calcium (about 700 mg/daily) whilst there are several reports indicating beneficial effects of calcium-rich diets. Aim of the preset study is to evaluate the effects of a low-sodium, low-lipid diet enriched in calcium, mainly from vegetables instead of dairy products, on blood pressure, body weight a main parameters of the glucose and lipid metabolisms.

This study is a randomized, parallel group trial that will be performed in the Outpatient Clinic. At least 150 patients with arterial hypertension and/or increased body weight (IMC> 28 kg/m2) will enter the study program. After a 3 month low-lipid low-salt diet that will be prescribed to all patients, they will be divided in two groups. The first will change the diet to that similar for total calories, percent composition of macronutrients and salt but enriched in calcium (about 1200 mg/daily) whilst the alternative group will continue the first diet. The observation period will be of 1 year with anthropometric (body weight and height, waist circumference), hemodynamic (blood pressure and heart rate) and metabolic (cholesterol, triglycerides, fasting blood glucose, uric acid, calcium, phosphorus, sodium and potassium) controls after 3-6 and 12 months.

DETAILED DESCRIPTION:
The DASH Study showed that the antihypertensive effects of a low-salt, low-lipid diet were significantly potentiated when the diet was enriched in calcium. This target may be reached either increasing the daily consumption of low-lipid milk and dairy products or increasing the daily consumption of calcium-rich vegetables.

In the Italian population the mean daily consumption of calcium is rather low, not exceeding 700 mg/daily whilst it would be desirable a daily consumption of 1200 mg/daily. Unfortunately there are in Italy very few dairy products (particularly low-lipid cheese) that would ensure a variable and palatable calcium-rich diet.

Aims of the present study are:

1. to prepare a low-sodium (about 3 g/daily) diet enrich in calcium (about 1200 mg/daily) and to compare the effects on blood pressure with those of a low-sodium diet similar to it in macronutrients but with a calcium content typical of the Mediterranean diet (no more than 700 mg/daily) (see Table 1);
2. to verify if this diet is able to improve the control of body weight and of the main parameters of the glucose and lipid metabolisms;
3. to evaluate if this diet is palatable enough to be prescribed in a long term study.

Patients:

At least 150 patients with arterial hypertension and/or overweight /obesity (IMC > 28 kg/m2) will be enrolled.

Methods:

1. evaluation of nutritional habits by an adequate frequency questionnaire at baseline, after a 3-month low-lipid low-sodium diet;
2. anthropometric measures (body weight, height, waist circumference);
3. measurements of blood pressure and heart rate;
4. measurements of serum total and HDL cholesterol serum triglycerides, fasting blood glucose, serum sodium potassium calcium and phosphorus.

Design of the study:

This is a randomized parallel-group study performed in the Outpatient Clinic. Patients enrolled in the study will be prescribed a low-sodium low-lipid diet for 3 months. At the end of the first phase they will be randomly divided in two groups:

1. Group A: patients will change their diet in a diet similar for total daily calories, sodium and macronutrients but enriched in calcium (1200 mg/daily) and will be followed up to 1 year with an intermediate control after the first 3 months;
2. Group B: patients will continue the low-lipid, low-sodium diet up to 1 year with an intermediate control after the first 3 months.

At baseline, after 3, 6 and 12 months of observation, patients will repeat the measurements 1-4 described in the Methods.

Composition in macro and micronutrients of the two diets

NUTRIENTS LOW-SODIUM DIET LOW-SODIUN CALCIUM- ENRICHED DIET PROTEINS (%) 17 17 LIPIDS (%) 27 28 SATURATED FATTY ACIDS (%) 7 7 MONOUNSATURATED (%) 16 17 POLTYUNSATURATED (%) 4 4 CHOLESTEROL ( mg) 132 140 CARBOHYDRATES (%) 56 54 SOLUBLE CHO (%) 18 17 FIBRE (g) 39 42 Na (mg) 1397 1377 K (mg) 3973 4067 Fe (mg) 16 21 Ca (mg) 650 1211 P (mg) 1285 1501

ELIGIBILITY:
Inclusion Criteria:

* age 30-70 years
* IMC >28 and < 35 kg/m2
* pharmacological treatment unchanged in the last 3 months

Exclusion Criteria:

* chronic kidney disease
* liver or chronic inflammatory bowel disease
* tumor

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Antihypertensive effects as measured by BP measurements | after 3-months of dietary treatment
  Measurements of blood pressure by sphygmomanometer.

SECONDARY OUTCOMES:
Effects on body weight as measured by scale | after 3-months of dietary treatment
  measurements of body weight
Effects on glucose metabolism as measured by fasting blood glucose | after 3 months of dietary treatment
  measurements of fasting blood glucose
Effects on lipid metabolism as measured by measurements of serum cholesterol, triglycerides and HDL-cholesterol | after 3 months of dietary treatment
  measurements of serum cholesterol, HDL-cholesterol, total triglycerides

OTHER OUTCOMES:
Long term feasibility of the diet as measured by adherence to dietary treatment | after 1 yearof dietary treatment
  to evaluate if this diet is palatable enough to be prescribed in a long term study by an appropriate questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Liberato Aldo Ferrara, MD, Principal Investigator — Dept. of Medicine and Surgery; Federico 2nd University of Naples
Locations (1):
- Hypertention Outpatient Clinic Dept. of Clinica Medica; Federico 2nd University of Naples, Naples, Naples, Italy